CLINICAL TRIAL: NCT05319769
Title: Non Fluoroscopic APpROach iN atriaL Fibrillation Ablation procEdureS
Acronym: APRONLESS
Status: Completed | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Matteo Bertini, Principal Investigator, University Hospital of Ferrara
Other Study IDs: 234/2022/Oss/AOUFe
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; ablation; radiofrequency; intracardiac echocardiography; zero fluoroscopy; arrhythmias
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Zero fluoroscopy: Zero fluoroscopy Patients undergoing AF ablation using the steerable introducer in combination with the 3D EAM system and intracardiac echocardiography.
  Reconstruction of a bipolar map of the right atrium with a mapping catheter. Then, the interatrial septum is reconstructed and the oval fossa is defined. Transseptal puncture is performed using the steerable introducer (which can be viewed on the EAM) through which, a transseptal needle is introduced. The introducer is positioned at the fossa ovalis. The transseptal needle is advanced to perform the puncture of the septum. After accessing the left atrium, the mapping catheter is introduced iusing the introducer, with which all the structures of the left atrium are mapped. In addition, with intracardiac echocardiography, it is possible to identify important structures such as the pulmonary veins and the esophagus. The pulmonary veins are isolated by means of a catheter.
  Interventions: Procedure: Atrial fibrillation ablation
- Traditional approach: Traditional approach Patients who have undergone atrial fibrillation ablation procedure using the traditional approach.
  The procedure is based on 3D reconstruction using intracardiac ultrasound first and then electroanatomical mapping of the left atrium through a transseptal approach guided by integration of fluoroscopy and intracardiac ultrasound. The transseptal puncture is performed using a transseptal needle which is brought into place using a long introducer with a dilator. The fluoroscopic support is essential as the introducer is not viewable with 3D mapping systems. After accessing the left atrium, through the previously used introducer, a mapping catheter is taken to the left atrium for electro-anatomical reconstruction. Subsequently, the antral pulmonary veins are isolated by means of an ablator catheter with irrigated tip.
  Interventions: Procedure: Atrial fibrillation ablation

INTERVENTIONS:
Procedure: Atrial fibrillation ablation — Pulmonary vein isolation

SUMMARY:
In electrophysiology, interventional procedures are often assisted by fluoroscopic guidance, exposing both patients and healthcare professionals to a considerable dose of radiation. Catheter ablation of atrial fibrillation has frequently involved the use of fluoroscopy: in fact, it incorporates greater complexity due to the need to perform the transseptal puncture.

A visible introducer in the 3D electro-anatomical mapping system (which does not involve the use of X-rays), has become an important tool for performing transseptal puncture: in particular, it is positioned at level of the oval fossa of the right atrium (puncture site); subsequently, the needle is introduced inside it; the intervention is guided both by electroanatomical mapping and by the use of intracardiac echocardiography for the identification of important anatomical landmarks.

The "zero rays" technique represents a valid alternative to fluoroscopic guidance, widely used and validated over the years. In fact, X-ray exposure in an atrial fibrillation ablation procedure can reach up to 60 mSv: the radiological risk makes it necessary to study safe and effective alternative techniques.

In this retrospective, observational and monocentric study, 50 catheter ablation procedures of atrial fibrillation will be examined, divided into two groups:

1. 25 patients who performed this procedure according to the classic approach, ie under fluoroscopic guidance;
2. 25 patients who performed this procedure using an ablative approach that involved the use of the introducer in combination with the 3D EAM system and intracardiac echocardiography.

Clinical efficacy will be assessed through a cardiological checkup and 24-hour electrocardiographic recording (ECG Holter) at 6 months.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common sustained adult tachyarrhythmia found in clinical practice. The prevalence of this arrhythmia in the general population varies from 2 to 4% and increases significantly in elderly patients and in carriers of diseases such as arterial hypertension, heart failure, coronary and valvular disease, obesity, diabetes mellitus and chronic kidney disease. In addition to being a marker of underlying heart or vascular disease, FA in itself is accompanied by an increased incidence of ischemic stroke, heart failure and dementia. The mechanisms underlying this arrhythmia are still debated, but seem to involve electrical and structural alterations of the atrium that constitute a morpho-functional substrate that facilitate its development.

Traditionally, five types of atrial fibrillation are distinguished, based on presentation, duration and term:

1. Newly diagnosed AF: first finding of AF, regardless of the duration, presence and severity of symptoms;
2. Paroxysmal AF: AF that resolves within seven days (spontaneously or through cardioversion);
3. Persistent AF: AF that lasts more than seven days or is cardioverted after seven days;
4. Long lasting AF: AF that lasts more than a year continuously, when a rhythm control strategy has been adopted.
5. Permanent AF: AF accepted by the patient (and by the attending physician) for which no further attempt to control the rhythm is undertaken.

Treatment include heart rate and / or rhythm control strategies, prevention of cerebral thromboembolism and reduction / elimination of symptoms, as well as control of major cardiovascular risk factors. The decision about the implementation of therapeutic strategies aimed at restoring and maintaining sinus rhythm must be shared between doctor and patient, weighing on the one hand the effect on quality of life and symptoms, and on the other the risk of toxic effects of drugs. used. When AF has been on for less than a year, an early rhythm control strategy has been shown to reduce the composite outcome of cardiovascular death, stroke, hospitalization for heart failure or acute coronary syndrome in the EAST-AFNET 4 clinical trial.

Trans catheter ablation is a well-established treatment for the reduction of AF relapses and is proposed in cases of paroxysmal and persistent AF. It is a procedure that consists in the antral circumferential disconnection of the pulmonary veins by radiofrequency, laser or cryoblation. It is a safe and effective technique for maintaining sinus rhythm and for improving symptoms. When antiarrhythmic drugs fail in rhythm control, the current ESC 2020 Guidelines place trans-catheter ablation in class I for paroxysmal and persistent AF with or without major risk factors for recurrence, while as a first therapeutic approach it is in class IIa for paroxysmal AF and IIb for persistent AF without major risk factors for relapse.

Advanced three-dimensional electro-anatomical mapping systems (3D EAM) have revolutionized the transcatheter ablative approach, allowing a new approach to the study of complex arrhythmias, such as FA. All the mapping systems, even if based on different principles, allow a precise localization of the scaler catheter, starting from the vascular access up to the heart chambers. While the catheter scans the different cardiac structures, the system records information about the catheter's position and uses the spatial and electrical data to create an accurate reproduction of the 3D geometry of the cardiac structures. All this has led to a reduction in the use of fluoroscopy and, in particular for the ablation of AF, there has been a reduction in radiation during these procedures even if a complete elimination has not yet been possible.

Intracardiac echocardiography is an imaging technique capable of visualizing heart structures in real time and with very high spatial resolution, as well as monitoring the position of the catheter within the heart chambers and quickly identifying any procedural complications, such as the formation of thrombus or pericardial effusion. A further advantage is represented by the reduction of the scan times. For these reasons, intracardiac echocardiography has largely replaced transesophageal echocardiography in many interventional procedures, including those of electrophysiology. In fact, intracardiac echocardiography allows the integration of images in real time with electro-anatomical mapping systems, allowing to map those structures that are not viewable under fluoroscopy, such as the atrial septum.

A bi-directional, deflectable guide introducer capable of being visualized on the 3D mapping system allows the visualization in real time, allowing to increase the efficiency during the mapping and positioning of the scaler catheter, reducing, up to zero, the scan times. It also has 2-degree bidirectional deflection capability, reaching up to 180 degrees in both directions.

Furthermore, it is extremely performing during the atrial septal puncture procedures: when, in fact, a dilator is introduced through introducer to perform the transseptal puncture, the presence of a smooth interface between the dilator and the tip of introducer allows access more easily to the left atrium, reducing the force required to advance the system through the atrial septum by 33%.

The fluoroscopic approach is widely validated and has represented for years the gold standard in electrophysiological study and ablation procedures. However, this approach exposes the operator and the patient to a high dose of radiation: in fact, during an AF ablation procedure, the radiological exposure can reach up to 60 mSv, thus increasing the absolute risk of developing lifetime cancer by 0.08%. It is therefore very necessary to apply the principles of ALARA (a slow as reasonably achievable) as established by the consent document of the American College of Cardiology of 1998.

Recently the trans catheter ablation procedures of AF have undergone a major increase. Considering, therefore, the wide diffusion of this technique and the high radiological exposure linked to the transseptal puncture and the isolation of the pulmonary veins, promoting an approach without radiological exposure becomes extremely crucial.

The rationale of this study is to evaluate the clinical and procedural features of an ablative approach using the steerable introducer in combination with the 3D EAM system and intracardiac echocardiography: the combination of these elements is potentially able to significantly reduce, to zero, the scanning times and to reduce procedural times, guaranteeing efficacy and safety. Complications will also be assessed at 30 days and the effectiveness of the procedure at six months.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal or persistent atrial fibrillation
* Atrial fibrillation ablation performed during study period
* Clinical follow-up and ECG-Holter recording during follow-up

Exclusion Criteria:

* Age < 18 years
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation (paroxysmal or persistent) treated with transcatheter ablation
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Fluoroscopy time | Intraprocedure
  Time of X-ray exposure
DAP | Intraprocedure
  Dose area product
Procedural time | Intraprocedure
  Total procedure time

SECONDARY OUTCOMES:
Time for PVI | Intraprocedure
  Pulmonary veins isolation time
Complications | 30 days
  Procedural complications, percardial effusion, groin hematoma, thromboembolism
Absence of atrial fibrillation recurrence | 6 months
  Freedom from new episodes of arrhythmias

CONTACTS AND LOCATIONS:
Locations (1):
- Matteo Bertini, Ferrara, Italy